CLINICAL TRIAL: NCT06483126
Title: The Benefits of Nature for Mood and Cognition in Persons With and Without Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Alice Cronin-Golomb, Director, Vision and Cognition Laboratory, Boston University Charles River Campus
Other Study IDs: 7175E
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease; Mood; Cognition
Keywords: Nature; Natural Environments
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Persons with Parkinson's disease (PwPD): Individuals with a diagnosis of Parkinson's disease
- Persons without Parkinson's disease: Healthy middle-aged and older adults

SUMMARY:
This online study aims to explore the benefits of nature for mood and cognition in persons with and without Parkinson's disease. For the purpose of this survey, "natural environment" refers to places that primarily consist of natural elements, such as vegetation, water bodies, and landscapes. This includes greenspaces (such as parks, gardens, neighborhood streets lined with trees, forests, or nature reserves) bluespaces (such as next to beaches, lakes, rivers, ponds, or waterfronts), and desert regions, among others.

DETAILED DESCRIPTION:
To participate in this online study, you will need an email address, and a smartphone or laptop/desktop with internet access. If you are eligible to participate, you will be sent a link to an online survey (Qualtrics). We will ask questions about demographic and health information, followed by questions about exercise habits, exposure to natural environments (including greenspaces and bluespaces, among others), and questionnaires assessing mood, motivation, cognition, sleep, stress, quality of life, and related functions. The survey should take roughly 20-25 minutes to complete. This is an observational study only, and not an interventional study.

Compensation: A $15 Amazon gift card will be offered to those who complete the survey all the way through with good effort.

ELIGIBILITY:
Inclusion Criteria:

For persons with Parkinson's disease:

* Participants must be at least 40 years old
* Have a diagnosis of idiopathic PD
* Be proficient English speakers
* Have functional vision
* Have internet access, and access to a smartphone/laptop/desktop

For persons without Parkinson's disease:

* Participants must be healthy middle-aged and older adults, with no diagnosis of neurological/neurodegenerative conditions
* Participants must be at least 40 years old
* Be proficient English speakers
* Have functional vision
* Have internet access, and access to a smartphone/laptop/desktop

Exclusion Criteria (both groups):

* Diagnosis of dementia
* Poor vision (non-functional range)
* Lack of access to internet or to a smartphone/ laptop/desktop computer.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with and without Parkinson's disease volunteering for an online study
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Nature Connection Index | Baseline
  Assesses the extent to which people feel connected to nature.
Perceived Restorativeness Scale | Baseline
  Assesses the extent to which particular environments have restorative qualities. Higher scores indicate greater perceived restorativeness.
Center for Epidemiological Studies Depression (CES-D) | Baseline
  Assesses depressive symptoms in the general population. Maximum score:60. Higher scores indicate more severe depression.
Parkinson's Disease Sleep Scale-2 | Baseline
  Assesses sleep and nocturnal disturbances in Parkinson's disease. Maximum score: 60. Higher scores indicate more frequent sleep disturbances.
Parkinson's Disease Questionnaire - 8 (PDQ-8) | Baseline
  Assesses Parkinson's disease-specific health-related quality of life. Maximum Score: 32. Higher scores indicate worse quality of life.
Perceived Stress Scale | Baseline
  Assesses how different situations affect feelings and perception of stress. Maximum score: 40. Higher scores indicate higher perceived stress.
NIH NeuroQoL measures | Baseline
  Assesses health-related quality of life in adults with neurological disorders. Higher scores on the sub-scales indicate worse outcomes.
Parkinson's Anxiety Scale (PAS) | Baseline
  Assesses the severity of anxiety symptoms in persons with Parkinson's disease. Maximum score:48. Higher scores indicate more severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Cronin-Golomb, PhD, Principal Investigator — Boston University
Locations (1):
- Vision and Cognition Laboratory, Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alcock I, White MP, Wheeler BW, Fleming LE, Depledge MH. Longitudinal effects on mental health of moving to greener and less green urban areas. Environ Sci Technol. 2014 Jan 21;48(2):1247-55. doi: 10.1021/es403688w. Epub 2014 Jan 7. PMID 24320055
- [Background] Gascon M, Triguero-Mas M, Martinez D, Dadvand P, Forns J, Plasencia A, Nieuwenhuijsen MJ. Mental health benefits of long-term exposure to residential green and blue spaces: a systematic review. Int J Environ Res Public Health. 2015 Apr 22;12(4):4354-79. doi: 10.3390/ijerph120404354. PMID 25913182
- [Background] Hartig T, Mitchell R, de Vries S, Frumkin H. Nature and health. Annu Rev Public Health. 2014;35:207-28. doi: 10.1146/annurev-publhealth-032013-182443. Epub 2014 Jan 2. PMID 24387090
- [Background] Rigolon A, Browning MHEM, McAnirlin O, Yoon HV. Green Space and Health Equity: A Systematic Review on the Potential of Green Space to Reduce Health Disparities. Int J Environ Res Public Health. 2021 Mar 4;18(5):2563. doi: 10.3390/ijerph18052563. PMID 33806546
- [Background] Rodriguez-Loureiro L, Casas L, Bauwelinck M, Lefebvre W, Vanpoucke C, Vanroelen C, Gadeyne S. Social inequalities in the associations between urban green spaces, self-perceived health and mortality in Brussels: Results from a census-based cohort study. Health Place. 2021 Jul;70:102603. doi: 10.1016/j.healthplace.2021.102603. Epub 2021 Jun 21. PMID 34166885
- [Background] Miller IN, Neargarder S, Risi MM, Cronin-Golomb A. Frontal and posterior subtypes of neuropsychological deficit in Parkinson's disease. Behav Neurosci. 2013 Apr;127(2):175-183. doi: 10.1037/a0031357. Epub 2013 Feb 11. PMID 23398433
- [Background] Cerin E, Barnett A, Shaw JE, Martino E, Knibbs LD, Tham R, Wheeler AJ, Anstey KJ. From urban neighbourhood environments to cognitive health: a cross-sectional analysis of the role of physical activity and sedentary behaviours. BMC Public Health. 2021 Dec 23;21(1):2320. doi: 10.1186/s12889-021-12375-3. PMID 34949175
- [Background] Cerin E, Barnett A, Shaw JE, Martino E, Knibbs LD, Tham R, Wheeler AJ, Anstey KJ. Urban Neighbourhood Environments, Cardiometabolic Health and Cognitive Function: A National Cross-Sectional Study of Middle-Aged and Older Adults in Australia. Toxics. 2022 Jan 7;10(1):23. doi: 10.3390/toxics10010023. PMID 35051065